CLINICAL TRIAL: NCT04044196
Title: Preoperative Psychological Risk Factors for the Retractable Capsulitis of the Shoulder After Shoulder Rotator Cuff Repair Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Clinical Research director, Hospital Ambroise Paré Paris
Other Study IDs: APR012018; 2018-A00148-47 (Other: ID-RCB)
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Frozen Shoulder; Rotator Cuff Tears
MeSH Terms: conditions — Bursitis; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Rotator cuff repair — Rotator cuff repair performed arthroscopically

SUMMARY:
The main objective of our study is to determine whether preoperative anxiety, depression and kinesiophobia are risk factors for retractile capsulitis after arthroscopic rotator cuff repair to best support these patients. patients postoperatively.

DETAILED DESCRIPTION:
The occurrence of a postoperative frozen shoulder after tendon repair of the rotator cuff of the shoulder is a devastating complication. It causes stiffness and slows down recovering. It associates a synovitis and a capsular retraction generating a transient but very incapacitating passive and active joint stiffness.

The evolution of capsulitis occurs in three phases:

* The first phase or cold phase is distinguished mainly by pain. The stiffness settles gradually. This phase lasts 2 to 9 months
* In the second phase or frozen phase lasting 4 to 12 months, the pain is less severe, but the rigidity is substantial.
* In the third phase, the function is gradually recovered and the pain disappears. This phase can last up to two years.

Some patients will get back full mobility of their shoulder in 12 to 18 months, while others may have persistent symptoms for several months.

The International Society of Arthroscopy, Knee Surgery and Orthopedic Sports Medicine recently codified the clinical diagnosis: active anterior elevation less than 100 °, external rotation elbow to body less than 10 °, internal rotation less than L5.

So if the diagnosis is better codified , prevention is the main concern. Some etiologies have been clearly identified. Systemic etiologies are reported: diabetes, thyroid pathologies, Dupuytren's disease and other factors such as ipsilateral breast surgery and myocardial infarction.

Psychological predispositions have long been suggested as risk factors for capsulitis, but a significant relationship has not been clearly established. The fear of having pain or an apathetic temperament could lead to a stay of the pains and curb the reeducation. In 1953, Coventry already evoked a "so called periarthritic personality" associating apathy, muscle contractures and a threshold of low pain. In 2014, De Beer investigated whether personality traits favored the occurrence of a retractable capsule primary or secondary to surgery but did not identify specific personality significantly more prone to stiffening of the shoulder.

Moreover, the fear of pain during movement or kinesiophobia and the avoidance behaviors generated are known factors in the persistence of pain and chronic limitations of function.

The main objective of our study is to determine whether preoperative anxiety, depression and kinesiophobia are risk factors for retractile capsulitis after arthroscopic rotator cuff repair to best support these patients. patients postoperatively.

Our hypothesis is that there is a psychological ground predisposing to the postoperative occurrence of a retractile capsulitis of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with rotator cuff rupture or subacromial conflict.
* Free and enlightened non-opposition

Exclusion Criteria:

* Pregnancy and breast feeding
* Associated repair of the scapular tendon
* Risk factors for capsulitis: diabetes, thyroid pathology, hypercholesterolemia, dupuytren's disease, homolateral breast surgery, history of myocardial infarction
* Patient not affiliated to a social security scheme
* Refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who undergo rotator cuff repair under arthroscopy
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
retractile capsulitis | 6 months postoperatively
  rate of patients with retractile capsulitis defined as active anterior elevation less than 100 °, external rotation elbow to body less than 10 °, internal rotation less than L5

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | preoperatively and 6 months after surgery
  self-questionnaire Scoring: Total score: Depression (D) and Anxiety (A) 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Tampa Scale for Kinesiophobia (TSK) | preoperatively and 6 months after surgery
  self-questionnaire The TSK consists of 17 questions. A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.
Numeric Pain Rating Scale | preoperatively and 6 months after surgery
  from "0" (no pain) to "10" (the worst pain)
Constant shoulder score | preoperatively and 6 months after surgery
  divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bauer, MD, PhD, Principal Investigator — Orthopaedic surgery department
Locations (2):
- France (2):
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Ambroise Paré Hospital, Boulogne-Billancourt, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aim F, Chevallier R, Marion B, Klouche S, Bastard C, Bauer T. Psychological risk factors for the occurrence of frozen shoulder after rotator cuff repair. Orthop Traumatol Surg Res. 2022 Apr;108(2):103212. doi: 10.1016/j.otsr.2022.103212. Epub 2022 Jan 22. PMID 35077897